CLINICAL TRIAL: NCT04159558
Title: Development and Evaluation of mHealth Solutions to Monitor and Involve Cardiometabolic Patients in Self-care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, José Joaquín Mira, University Professor with a related position as Clinical Psychologist in SNS, Universidad Miguel Hernandez de Elche
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18/324
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Hypertension; Diabetes; Heart Failure; Copd; Asthma; Obesity
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Heart Failure; Pulmonary Disease, Chronic Obstructive; Asthma; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- experimental hypertension (Experimental): The subjects with Hypertension will be trained in the use of the personalized help tool and will use it during a period of 3 months.
  Interventions: Device: Mobile application
- experimental diabetes (Experimental): The subjects with Diabetes will be trained in the use of the personalized help tool and will use it during a period of 3 months.
  Interventions: Device: Mobile application
- experimental heart failure (Experimental): The subjects with Heart failure will be trained in the use of the personalized help tool and will use it during a period of 3 months.
  Interventions: Device: Mobile application
- experimental copd (Experimental): The subjects with COPD will be trained in the use of the personalized help tool and will use it during a period of 3 months.
  Interventions: Device: Mobile application
- experimental asthma (Experimental): The subjects with Asthma will be trained in the use of the personalized help tool and will use it during a period of 3 months.
  Interventions: Device: Mobile application
- experimental obesity (Experimental): The subjects with Obesity will be trained in the use of the personalized help tool and will use it during a period of 3 months.
  Interventions: Device: Mobile application

INTERVENTIONS:
Device: Mobile application — Experimental group will use a mobile application to help them in their self-care

SUMMARY:
To develop, using barcode systems and virtual pillbox (TuMedicina and Alice), an App aimed at patients and carers of patients with cardiometabolic diseases as the main diagnosis, over 45 years of age, who have one or more pathologies and use one or more drugs on a daily basis and to analyze their effectiveness in terms of achieving therapeutic objectives, self-efficacy and self-efficacy in self-care or provision of care (as the case may be), healthy behavior, therapeutic compliance and safe use of medication.

DETAILED DESCRIPTION:
In order to achieve the objective of this study, an experimental study will carry out on patients with cardiometabolic and respiratory diseases and their caregivers. A participation of 100 patients and 85 caregivers is planned. The aim is for them to use the mobile application developed over three months in order to evaluate their health improvement comparing several clinical and analytic parameters before and after the use of the App, and also evaluating the satisfaction of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Cardio-metabolic disease, respiratory disease or neurologic disease

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-04-24 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with the mobile application assessed by an ad hoc questionnaire | 3 months
  % of participants who were satisfied with the mobile application assessed by an ad hoc questionnaire

SECONDARY OUTCOMES:
Treatment adherence assessed by Morisky Medication Adherence Scale (MMAS) | 3 months
  % of participants who improve their treatment adherence assessed by Morisky Medication Adherence Scale (MMAS)

OTHER OUTCOMES:
Health goals compliance assessed by an ad hoc questionnaire | 3 months
  % of participants who compliance their health goals assessed by an ad hoc questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Miguel Hernández University, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No